CLINICAL TRIAL: NCT00548912
Title: Cardiac Magnetic Resonance Imaging in Hemodialysis Patients
Brief Title: Left Ventricular Hypertrophy and Spironolactone in End Stage Renal Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study ended
Sponsor: Dawnmarie DeFazio (Other)
Responsible Party: Sponsor-Investigator, Dawnmarie DeFazio, Nephrolgist, Co-Investigator, West Penn Allegheny Health System
Organization: West Penn Allegheny Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC-3267
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Hemodialysis; Spironolactone
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Spironolactone

ARMS (1):
- 1 group - no arms (Other): no arm just error message
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone

SUMMARY:
The hypothesis of this trial is to assess the effect of spironolactone on heart size and mass

DETAILED DESCRIPTION:
Dialysis patients have significant morbidity and mortality associated with left ventricular hypertrophy and cardiac failure. Aldosterone may have an important role in the development of myocardial hypertrophy and remodeling. Animal studies have demonstrated beneficial effects of aldosterone antagonists on myocardial hypertrophy, and human studies have shown significant survival benefit in a non-dialysis population with congestive heart failure. This study evaluates the effect of spironolactone (an aldosterone receptor antagonist) on cardiac hypertrophy in the end-stage renal disease population.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients

Exclusion Criteria:

* non compliance
* hyperkalemia
* pregnancy
* expected survival less than 9 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marcus, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States